CLINICAL TRIAL: NCT00350506
Title: An Open-label, Non-randomized, Multi-center Trial Evaluating the Clinical Applicability, Correlation, and Modeling of Cardiac CT Using 64 Detector Row VCT
Brief Title: A Trial Evaluating the Clinical Applicability, Correlation, and Modeling of Cardiac CT Using 64 Detector Row VCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision (due to low subject enrollment)
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VCT-001
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- 64 Channel VCT (Experimental): All subjects underwent Coronary Computed Tomographic Angiography (CCTA) after receiving an intravenous (IV) administration of Visipaque (320 mgI/mL), to be followed by catheter coronary angiography (CATH).
  Interventions: Device: 64 Channel VCT

INTERVENTIONS:
Device: 64 Channel VCT

SUMMARY:
To compare computed tomography (CT) images (pictures) of the coronary arteries using the General Electric (GE) LightSpeed VCT scanner with x-ray coronary angiography in patients referred for an x-ray coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective diagnostic catheterization OR
* Elective diagnostic catheterization has been performed within the past 2 weeks but no less than 24 hours prior to the coronary CTA procedure with no intervention performed or change of the patient clinical status.
* Age ≥18 years but ≤75 years.

Exclusion Criteria:

* Prior coronary stent implantation
* Prior coronary artery bypass grafting or other heart surgery
* Prior pacemaker or internal defibrillator lead implantation
* Prior artificial heart valve
* Biochemical renal insufficiency (CrSerum > 1.6) or on dialysis
* Resting HR > 100 at the time of enrollment
* Contraindication to β-blockade or calcium channel blocker

  * NYHA-IV
  * High-grade atrioventricular (AV) block
  * Systolic blood pressure <90 mm Hg
  * Severe asthma or active bronchospasm and/or chronic obstructive pulmonary disease
* Atrial fibrillation
* Inability to provide informed consent
* Evidence of ongoing or active clinical instability

  * Acute chest pain (sudden onset)
  * Acute myocardial infarction
  * Cardiac shock
  * Acute pulmonary edema

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Centofanti, MS, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States